CLINICAL TRIAL: NCT01328496
Title: Umbilical Cord Blood Transplantation In Patients With Hematologic Malignancies Using A Myeloablative Preparative Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: The Hartwell Foundation (Other); Assisi Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCBT01; NCI-2011-03700 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-03

CONDITIONS: Hematologic Malignancies; Disorder Related to Transplantation; Hematopoietic Malignancy
Keywords: Hematologic Malignancies; Umbilical Cord Blood transplantation; Hematopoietic Cell Transplantation
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Research Arm (Other): Participant with high-risk hematologic malignancies undergoing Hematopoietic Cell Transplantation, who do not have a suitable Human Leukocyte Antigen -matched related/sibling donor, Matched Unrelated Donor or Killer immunoglobulin receptors ligand mismatched haploidentical donor identified, will receive a single UCB unit.
  Intervention: Preparative Regimen
  Interventions: Drug: Preparative Regimen
- Observation Arm (Other): Patients requiring two UCB units will be eligible for UCBT01 on the observational arm.
  Intervention: Preparative Regimen
  Interventions: Drug: Preparative Regimen

INTERVENTIONS:
Drug: Preparative Regimen — Fludarabine (75 mg/m2), fractionated total body irradiation (TBI) (12.0 Gy), and cyclophosphamide (120mg/kg) with mesna. Fludarabine will be given once a day at 25 mg/m2 for three days on day -10 to day -8, TBI will be given twice a day at 150 cGy for four days on day -7 to day -4, and cyclophosphamide will be given once a day for at 60mg/kg for two days on day -3 and day -2.
  Post-transplantation immunosuppression with cyclosporine and MMF will begin on day -3. Cord Blood infusion will occur on day 0 and G-CSF will start on day +1.

SUMMARY:
In this study, participants with high-risk hematologic malignancies undergoing hematopoietic cell transplantation (HCT), who do not have a suitable human leukocyte antigen (HLA)-matched related/sibling donor (MSD), matched unrelated donor (MURD) or killer-immunoglobulin receptors (KIR) ligand mismatched haploidentical donor identified, will receive an umbilical cord blood transplantation (UCBT) using a myeloablative preparative regimen.

The preparative regimen includes fludarabine (75 mg/m2), fractionated total body irradiation (TBI) (10.0 Gy), and cyclophosphamide (120mg/kg) with mesna. Fludarabine will be given once a day at 25 mg/m2 for three days on day -10 to day -8, TBI will be given twice a day at 150 cGy for four days on day -7 to day -4, and cyclophosphamide will be given once a day for at 60mg/kg for two days on day -3 and day -2. Post-transplantation immunosuppression with cyclosporine and MMF will begin on day -3. Cord Blood infusion will occur on day 0 and G-CSF will start on day +1.

DETAILED DESCRIPTION:
The primary objectives is to estimate the event-free survival (EFS) at one-year post-transplant for research participants with high-risk hematologic malignancies undergoing hematopoietic cell transplantation (HCT) using single unit umbilical cord blood (UCB).

Secondary objectives are:

* Describe the clinical outcome of patients undergoing a double unit UCBT.
* Estimate the incidence and severity of acute and chronic graft versus host disease (GVHD) of patients enrolled in the research arm.
* Estimate the incidence and time to neutrophil and platelet engraftment among patients enrolled in the research arm.
* Estimate the incidence of transplant related mortality (TRM) and transplant related morbidity in the first 100 days after transplantation among patients enrolled in the research

Exploratory Objectives are:

* Assess the relationship between pre-transplant minimal residual disease (MRD) with transplant outcomes.
* Record immune reconstitution parameters, including chimerism analysis, quantitative lymphocyte subsets, T cell receptor excision circle (TREC) and spectratyping. Immunophenotyping and functional assays of T, B and NK cells and lymphocytes will also be evaluated.
* Evaluate the determinants of engraftment.

ELIGIBILITY:
Inclusion Criteria:

* Age less than or equal to 21 years old.
* Has a partially HLA-matched single or double UCB product
* High-risk hematologic malignancy.
* High risk ALL in CR1, ALL in High risk CR2, ALL in CR3 or subsequent.
* AML in high risk CR1, AML in CR2 or subsequent
* AML in first relapse with < 25% blasts in BM
* Therapy related AML, with prior malignancy in CR > 12mo
* MDS, primary or secondary
* NK cell, biphenotypic, or undifferentiated leukemia in CR1 or subsequent.
* CML in accelerated phase, or in chronic phase with persistent molecular positivity or intolerance to tyrosine kinase inhibitor.
* Hodgkin lymphoma in CR2 or subsequent after failure of prior autologous HCT, or unable to mobilize stem cells for autologous HCT.
* Non-Hodgkin lymphoma in CR2 or subsequent after failure of prior autologous HCT, or unable to mobilize stem cells for autologous HCT.
* JMML
* All patients with evidence of CNS leukemia must be treated and be in CNS CR to be eligible for study.

Patient must fulfill pre-transplant evaluation:

* Cardiac shortening fraction ≥ 26%.
* Creatinine clearance ≥ 70 ml/min/1.73m2.
* Forced vital capacity (FVC) ≥ 50% of predicted value or pulse oximetry ≥ 92% on room air.
* Karnofsky (≥ 16 years) or Lansky (<16 years) performance score ≥ 70
* Bilirubin ≤ 2.5 mg/dL.
* Alanine aminotransferase (ALT) ≤ 5 times the upper limit of normal for age.
* Aspartate aminotransferase (AST) ≤ 5 times the upper limit of normal for age.

Exclusion Criteria:

* Patient has a suitable MSD, volunteer MURD, or KIR mismatched haploidentical donor available in the necessary time for stem cell donation.
* Patient has any other active malignancy other than the one for which HCT is indicated.
* Patient had a prior allogeneic HCT
* Patient had an autologous HCT within the previous 12 months.
* Patient is pregnant as confirmed by positive serum or urine pregnancy test within 14 days prior to enrollment.
* Patient is lactating
* Patient has Down Syndrome
* Patient has a current uncontrolled bacterial, fungal, or viral infection per the judgment of the PI.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2011-06-15 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amr Qudeimat, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fourteen patients were enrolled at St. Jude Children's Research Hospital between September 2011 and April 2014.
Groups:
- Research Arm: Participant with high-risk hematologic malignancies undergoing Hematopoietic Cell Transplantation, who do not have a suitable Human Leukocyte Antigen -matched related/sibling donor, Matched Unrelated Donor or Killer immunoglobulin receptors ligand mismatched haploidentical donor identified, will receive a single UCB unit.
  Intervention: Preparative Regimen
  Preparative Regimen: Fludarabine (75 mg/m2), fractionated total body irradiation (TBI) (12.0 Gy), and cyclophosphamide (120mg/kg) with mesna. Fludarabine will be given once a day at 25 mg/m2 for three days on day -10 to day -8, TBI will be given twice a day at 150 cGy for four days on day -7 to day -4, and cyclophosphamide will be given once a day for at 60mg/kg for two days on day -3 and day -2.
  Post-transplantation immunosuppression with cyclosporine and MMF will begin on day -3. Cord Blood infusion will occur on day 0 and G-CSF will start on day +1.
- Observational Arm: Patients requiring two UCB units will be eligible for UCBT01 on the observational arm.
  Intervention: Preparative Regimen
  Preparative Regimen: Fludarabine (75 mg/m2), fractionated total body irradiation (TBI) (12.0 Gy), and cyclophosphamide (120mg/kg) with mesna. Fludarabine will be given once a day at 25 mg/m2 for three days on day -10 to day -8, TBI will be given twice a day at 150 cGy for four days on day -7 to day -4, and cyclophosphamide will be given once a day for at 60mg/kg for two days on day -3 and day -2.
  Post-transplantation immunosuppression with cyclosporine and MMF will begin on day -3. Cord Blood infusion will occur on day 0 and G-CSF will start on day +1.
Period: Overall Study
Arm/Group | Research Arm | Observational Arm
Started | 10 | 4
Completed | 9 | 4
Not Completed | 1 | 0
Not completed — Significant Change in Health Status | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Research Arm | Observational Arm | Total
Number analyzed (Participants) | 9 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.40 (2.54) | 14.3 (2.98) | 6.76 (5.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Mexican/Chicano | 1 | 0 | 1
  NOS Spanish, Hispanic, latino | 2 | 2 | 4
  Non Spanish speaking, Non Hispanic | 3 | 2 | 5
  Puerto Rican | 2 | 0 | 2
  Declined to respond | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival (EFS) for Research Participants
Description: Estimate EFS for research participants at one-year post transplant by using single unit umbilical cord blood. The event is defined as relapse, graft failure, death due to any cause. The number of participants who did not experience any of those events (relapse, graft failure, death due to any cause) at year 1 post-transplant was given.
Time Frame: 1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Research Arm
Number analyzed (Participants) | 9
Participants | 4

2. Secondary Outcome: Number of Observational Arm Participants Engrafted
Description: For patients enrolled in the observational arm (undergoing a double unit UCBT), the number of patients engrafted was given.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Observational Arm
Number analyzed (Participants) | 4
Participants | 3

3. Secondary Outcome: Number of Observational Arm Patients Who Relapsed
Description: The number of observational arm patients who relapsed was given.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Observational Arm
Number analyzed (Participants) | 4
Participants | 1

4. Secondary Outcome: Number of Deaths of Observational Arm Patients
Description: The number of observational arm patients who died was given.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Observational Arm
Number analyzed (Participants) | 4
Participants | 2

5. Secondary Outcome: Number of Observational Arm Patients With Transplant-related Mortality (TRM)
Description: The number of patients with TRM within the first 100 days post transplant was given.
Time Frame: First 100 days
Measure: Count of Participants; unit: Participants
Groups:
- Observational Arm: Patients requiring two UCB units will be eligible for UCBT01 on the observationalal arm.
  Intervention: Preparative Regimen
  Preparative Regimen: Fludarabine (75 mg/m2), fractionated total body irradiation (TBI) (12.0 Gy), and cyclophosphamide (120mg/kg) with mesna. Fludarabine will be given once a day at 25 mg/m2 for three days on day -10 to day -8, TBI will be given twice a day at 150 cGy for four days on day -7 to day -4, and cyclophosphamide will be given once a day for at 60mg/kg for two days on day -3 and day -2.
  Post-transplantation immunosuppression with cyclosporine and MMF will begin on day -3. Cord Blood infusion will occur on day 0 and G-CSF will start on day +1.
Arm/Group | Observational Arm
Number analyzed (Participants) | 4
Participants | 1

6. Secondary Outcome: Number of Participants With Acute GVHD
Description: The number of participants with incidence of acute GVHD by grade was given. Participants are graded on a scale from 1 to 4, with 1 being mild and 4 being severe.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Research Arm | Observational Arm
Number analyzed (Participants) | 9 | 4
Participants
  Grade 1 | 2 | 0
  Grade 2 | 1 | 0
  Grade 3 | 1 | 1
  Grade 4 | 0 | 0
  No Acute GVHD | 5 | 3

7. Secondary Outcome: Number of Participants With Chronic GVHD
Description: Due to the small sample size, cumulative incidence analysis was not done. The incidence of chronic GVHD was evaluated using NIH Consensus Global Severity Scoring. The number of patients with incidence of chronic GVHD by severity was provided.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Research Arm | Observational Arm
Number analyzed (Participants) | 9 | 4
Participants
  Mild | 0 | 0
  Moderate | 0 | 0
  Severe | 0 | 0
  No Chronic GVHD | 9 | 4

8. Secondary Outcome: Time to Engraftment of Research Arm Participants
Description: Platelet engraftment was defined as platelet count ≥20,000/mm^3 for 3 consecutive tests performed on different days with no platelet transfusions in the preceding 7 days. Neutrophil engraftment will be defined as achieving ANC ≥ 500/mm3 for 3 consecutive tests performed on different days with evidence of donor cell engraftment. Descriptive statistics are provided.
Time Frame: first 100 days post transplant
Population: Those patients who did not reach engraftment are not included in the results provided below.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Research Arm
Number analyzed (Participants) | 9
Days
  Days to Platelets ≥20,000: number analyzed (Participants) | 6
  Days to Platelets ≥20,000 | 42.67 (8.80)
  Days to ANC ≥500 | 17.11 (5.93)

9. Secondary Outcome: Incidence of Transplant-related Mortality (TRM)
Description: TRM is death occurring in patients in continuous complete remission. The numbers of patients with TRM was given.
Time Frame: first 100 days post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Research Arm | Observational Arm
Number analyzed (Participants) | 9 | 4
Participants | 0 | 1

10. Secondary Outcome: The Number of Participants With Transplant-related Morbidity
Description: Any patient who had adverse events listed either as probable or definite in the first 100 days post-transplant are counted as transplant related morbidity. The number of patients with transplant-related morbidity was given.
Time Frame: first 100 days post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Research Arm | Observational Arm
Number analyzed (Participants) | 9 | 4
Participants | 8 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout from the start of initiation of conditioning to one year post transplant.
Groups:
- Observation Arm: Patients requiring two UCB units will be eligible for UCBT01 on the observational arm.
  Intervention: Preparative Regimen
  Preparative Regimen: Fludarabine (75 mg/m2), fractionated total body irradiation (TBI) (12.0 Gy), and cyclophosphamide (120mg/kg) with mesna. Fludarabine will be given once a day at 25 mg/m2 for three days on day -10 to day -8, TBI will be given twice a day at 150 cGy for four days on day -7 to day -4, and cyclophosphamide will be given once a day for at 60mg/kg for two days on day -3 and day -2.
  Post-transplantation immunosuppression with cyclosporine and MMF will begin on day -3. Cord Blood infusion will occur on day 0 and G-CSF will start on day +1.
Arm/Group | Research Arm | Observation Arm
All-Cause Mortality (participants affected / at risk) | 4/9 | 2/4
Serious Adverse Events (participants affected / at risk) | 7/9 | 3/4
Other Adverse Events (participants affected / at risk) | 9/9 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Research Arm (N=9) | Observation Arm (N=4)
Anemia, Hemolytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Effusion, Pericardial (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (disorder) (Cardiac disorders) | 1 (1) | 0 (0)
Fever without neutropenia (General disorders) | 5 (14) | 3 (3)
Dehydration (disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Infection, coagulase negative staph, blood (Infections and infestations) | 1 (1) | 0 (0)
Infection, enterococcus faecalis, blood (Infections and infestations) | 1 (1) | 0 (0)
Infection, escherichia coli, blood (Infections and infestations) | 1 (2) | 0 (0)
Infection, escherichia coli, urine (Infections and infestations) | 1 (1) | 0 (0)
Hyperkalemia (disorder) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute respiratory distress (finding) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Left pneumothorax (disorder) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Right pneumothorax (disorder) (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Effusion, pericardial (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (PRES) (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Research Arm (N=9) | Observation Arm (N=4)
Anemia, hemolytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Edema, generalized (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Edema, lower extremity (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (9) | 3 (3)
Febrile neutropenia (disorder) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2)
Fever without neutropenia (Cardiac disorders) | 2 (3) | 0 (0)
Hypertension (Cardiac disorders) | 7 (7) | 2 (2)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 3 (4)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (disorder) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis, oral mucosa (Gastrointestinal disorders) | 2 (2) | 0 (0)
vomiting (disorder) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever without neutropenia (General disorders) | 0 (0) | 1 (1)
Veno-occlusive disease, hepatic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Acute infusion reaction, acetaminophen (Immune system disorders) | 0 (0) | 1 (1)
Acute infusion reaction, stem cells (Immune system disorders) | 0 (0) | 1 (1)
Engraftment syndrome (Immune system disorders) | 2 (2) | 1 (1)
Adenoviral enteritis (disorder) (Infections and infestations) | 0 (0) | 1 (1)
CMV reactivation (Infections and infestations) | 0 (0) | 1 (1)
Enteritis (Infections and infestations) | 0 (0) | 1 (1)
Infection, adenovirus, blood (Infections and infestations) | 0 (0) | 1 (1)
Infection, adenovirus, stool (Infections and infestations) | 3 (3) | 2 (2)
Infection, aspergillus, lung (Infections and infestations) | 0 (0) | 1 (1)
Infection, BK virus, blood (Infections and infestations) | 1 (1) | 1 (1)
Infection, BK virus, urine (Infections and infestations) | 2 (9) | 1 (2)
Infection, clostridium difficile, stool (Infections and infestations) | 3 (3) | 1 (1)
Infection, enterococcus faecium, vancomycin resistant, blood (Infections and infestations) | 0 (0) | 1 (1)
Infection, enterococcus faecium, vancomycin resistant, bronchus (Infections and infestations) | 0 (0) | 1 (1)
Infection, enterococcus faecium, vancomycin resistant, penis (Infections and infestations) | 0 (0) | 1 (1)
Infection, enterocuccus faecium, vancomycin resistant, urine (Infections and infestations) | 0 (0) | 1 (1)
Infection, gram positive cocci (Infections and infestations) | 0 (0) | 1 (1)
Infection, human herpes virus 6 (Infections and infestations) | 0 (0) | 2 (2)
Infection, human herpes virus 6, blood (Infections and infestations) | 6 (6) | 1 (1)
Infection, human herpes virus 6, cerebrospinal fluid (Infections and infestations) | 0 (0) | 1 (1)
Infection, influenza B, nasal (Infections and infestations) | 0 (0) | 1 (1)
Infection, rotavirus, stool (Infections and infestations) | 2 (2) | 1 (1)
Infection, staphylococcus, urine (Infections and infestations) | 1 (1) | 1 (1)
Infection, streptococcus viridans, blood (Infections and infestations) | 0 (0) | 1 (1)
Tinea capitis (Infections and infestations) | 0 (0) | 1 (1)
Infection, adenovirus, nasal (Infections and infestations) | 1 (1) | 0 (0)
Infection, candida albicans (Infections and infestations) | 1 (2) | 0 (0)
Infection, enterobacter cloacae complex, Hickman Line (Infections and infestations) | 1 (1) | 0 (0)
Infection, enterobacter cloacae, blood (Infections and infestations) | 1 (2) | 0 (0)
Infection, herpes simplex virus, blood (Infections and infestations) | 1 (1) | 0 (0)
Infection, herpes simplex virus, oral mucosa (Infections and infestations) | 1 (1) | 0 (0)
Infection, herpes simplex, lip (Infections and infestations) | 1 (1) | 0 (0)
Infection, klebsiella oxytoca, blood (Infections and infestations) | 1 (1) | 0 (0)
Infection, klebsiella pneumoniae, blood (Infections and infestations) | 1 (1) | 0 (0)
Infection, pseudomonas aeruginosa, blood (Infections and infestations) | 1 (1) | 0 (0)
Infection, pseudomonas aeruginosa, rectum (Infections and infestations) | 1 (1) | 0 (0)
Infection, pseudomonas, tracheal aspirate (Infections and infestations) | 1 (1) | 0 (0)
Infection, sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Infection, staphylococcus aureus, blood (Infections and infestations) | 2 (2) | 0 (0)
Infection, staphylococcus aureus, Hickman Line (Infections and infestations) | 1 (1) | 0 (0)
Infection, staphylococcus, coagulase positive (Infections and infestations) | 1 (1) | 0 (0)
Infection, stenotrophomonas maltophilia, CVAD (Infections and infestations) | 1 (1) | 0 (0)
Infection, vancomycin resistant enterococcus (Infections and infestations) | 1 (1) | 0 (0)
Infection, vancomycin resistant enterococcus faecium, stool (Infections and infestations) | 1 (2) | 0 (0)
Infection, vancomycin resistant enterococcus, rectum (Infections and infestations) | 1 (2) | 0 (0)
Respiratory syncytial virus (RSV) (Infections and infestations) | 1 (1) | 0 (0)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypocalcemia (disorder) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesemia (disorder) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Demyelination (morphologic abnormality) (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy, motor (Nervous system disorders) | 0 (0) | 1 (1)
Syndenham's chorea (Nervous system disorders) | 1 (1) | 0 (0)
Mood alteration-anxiety/agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Severe depression (disorder) (Psychiatric disorders) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis, hemorrhagic (Renal and urinary disorders) | 1 (1) | 3 (3)
Failure, renal (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchiolitis obliterans organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Infiltrates, pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Lesion of lung (finding) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion, left (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia, middle lobe, right (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary nodules, consistent with fungal disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rash, generalized (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes